CLINICAL TRIAL: NCT03838848
Title: A Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of KN046 in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: KN046 in Patients With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cohort A,B,C end enrollments. Cohort D and E were considered to have no significant clinical benefit at the SMC meeting and decided to terminate enrollment.
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN046-201
Record Dates: First submitted 2019-02-01; First posted 2019-02-12 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Cohort A, B and C are carried out in sequence, a Scientific Monitoring Committee (SMC) will decide whether to enter the next group (A to B, B to C).
  Cohort D: 1L NSCLC (EGFR-sensitive mutation (Ex19del or L858R), progression after at least one line treatemtn of EGFR TKIs, and no prior systemic platinum-containing chemotherapy); Cohort E: ≥ 2L NSCLC (failure or intolerance of 1L platinum-doublet chemotherapy; and failure of PD-1/PD-L1 checkpoint inhibitor therapy);
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): Subjects with Non-small Cell Lung Cancer (NSCLC) (failed or did not tolerant to platinum-containing regime and did not treat with programmed cell death protein 1/the programmed death-ligand 1 (PD1/PDL-1) checkpoint inhibitor previously) will receive KN046 3 milligram per kilogram (mg/kg), every other weeks (Q2W)
  Interventions: Drug: KN046
- Cohort B (Experimental): Subjects with NSCLC (failed or did not tolerant to platinum-containing regime and did not treat with PD1/PDL-1 checkpoint inhibitor previously) will receive KN046 5 mg/kg, Q2W
  Interventions: Drug: KN046
- Cohort C (Experimental): Subjects with NSCLC (failed or did not tolerant to platinum-containing regime and failed to PD1/PDL-1 checkpoint inhibitor) will receive KN046
  Interventions: Drug: KN046
- Cohort D (Experimental): 1L NSCLC (EGFR-sensitive mutation (Ex19del or L858R), progression after at least one line treatemtn of EGFR TKIs, and no prior systemic platinum-containing chemotherapy), will receive KN046 5 mg/kg Q3W in combination with pemetrexed and carboplatin
  Interventions: Drug: KN046; Drug: Carboplatin; Drug: Pemetrexed
- Cohort E (Experimental): ≥ 2L NSCLC (failure or intolerance of 1L platinum-doublet chemotherapy; and failure of PD-1/PD-L1 checkpoint inhibitor therapy), will receive KN046 in combination with ningetinib
  Interventions: Drug: KN046; Drug: Ningetinib

INTERVENTIONS:
Drug: KN046 — 3mg/kg, Q2W, intravenous injection (IV)
  Other Names: Recombinant Humanized PD-L1/CTLA-4 Bispecific Single Domain Antibody Fc Fusion Protein Injection
  Arms: Cohort A
Drug: KN046 — 5mg/kg, Q2W, intravenous injection (IV)
  Other Names: Recombinant Humanized PD-L1/CTLA-4 Bispecific Single Domain Antibody Fc Fusion Protein Injection
  Arms: Cohort B; Cohort C; Cohort E
Drug: KN046 — 5mg/kg, Q3W, intravenous injection (IV)
  Other Names: Recombinant Humanized PD-L1/CTLA-4 Bispecific Single Domain Antibody Fc Fusion Protein Injection
  Arms: Cohort D
Drug: Carboplatin — AUC 5 IV Q3W; total dose calculated according to the Calvert formula, with the highest dose not exceeding 750 mg; 4 cycles.
  Arms: Cohort D
Drug: Pemetrexed — 500 mg/m2, Q3W, intravenous injection (IV)
  Arms: Cohort D
Drug: Ningetinib — Oral, QD
  Arms: Cohort E

SUMMARY:
This is a phase II, open label, multicenter study in subjects with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
A Phase 2 Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of KN046 in Subjects with Advanced Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent form(ICF);
2. Age ≥ 18 years and ≤ 75 years, male or female;
3. Histologically or cytologically documented NSCLC,Stage IV (AJCC Version 8) .
4. At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1;
5. Biopsy specimens obtained from nonradiated areas within 1 year, formalin-fixed, paraffin-embedded blocks containing tumor tissues suitable for biomarker determination, or 15-20 slides (more slides are encouraged to be provided with a minimum of 8 slides; if less than 8 slides are provided, the subject may also be enrolled after consultation and agreement between the Sponsor and the investigator); and fresh biopsy samples collected within 42 days prior to the first dose are required for determination in Cohorts C, D, and E;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Life expectancy > 12 weeks;
8. Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
9. Ability to comply with treatment, procedures and pharmacokinetics (PK) sample collection and the required study follow-up procedures

Exclusion Criteria:

1. Known brain metastasis or another Central Nervous System (CNS) metastasis that is either symptomatic or untreated.
2. Having participated in any interventional clinical study within 28 days prior to drug administration in this study.
3. Having received other anti-tumor therapy within 28 days before administration in this study, including traditional Chinese medicine with anti-tumor indications;
4. Having received major surgical treatment (such as major abdominal, transthoracic surgery; excluding diagnostic aspiration or peripheral vascular access replacement) within 28 days prior to drug administration in this study;
5. Having received radical radiotherapy within 3 months prior to drug administration in this study; palliative radiation therapy within 2 weeks prior to the first dose is allowed, the radiation dose meets the diagnostic and treatment criteria for local palliative treatment, and the radiation coverage is less than 30% of the bone marrow area;
6. Subjects who require systemic corticosteroids (≥ 10 mg/day prednisone or equivalent dose of other corticosteroids) or immunosuppressive therapy within 14 days prior to drug administration in this study; except for inhaled or topical corticosteroids, or physiologic replacement doses of corticosteroids for adrenal insufficiency; short-term (≤ 7 days) corticosteroids are allowed for prophylaxis (e.g., contrast media allergy) or for the treatment of non-autoimmune disorders (e.g., delayed type hypersensitivity due to contact allergens);
7. Having received live vaccines (including live attenuated vaccines) within 28 days prior to drug administration in this study;
8. Previous or current interstitial pneumonia/pneumopathy; Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded.
9. Subjects who have prior or current autoimmune diseases;
10. Subjects who have other malignancies within 5 years before the first dose;
11. Active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection, Known HIV infection or known history of acquired immune deficient syndrome (AIDS).
12. Any unresolved the Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2 toxicities from prior anti-cancer therapy except for vitiligo, alopecia;
13. History of allogeneic bone marrow or organ transplantation;
14. Prior history of allergic reaction, hypersensitivity reaction, and intolerance to antibody drugs; history of significant allergy to drugs;
15. Pregnant and/or lactating women;
16. Other conditions that, in the opinion of the investigator, will affect the safety or compliance of the subjects with the study treatment, including but not limited to psychiatric disorders, uncontrolled moderate to severe serous cavity effusions with large amounts of serous cavity effusions or requiring repeated drainage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
ORR | 2 years
  clinical response rate (ORR) as determined by the independent review board (IRC) based on RECIST 1.1 criteria
DOR | 2 years
  clinical response time (DOR) as determined by the independent review board (IRC) based on RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong A, Li W, Li X, Fan Y, Ma Z, Fang J, Xie Q, Zhuang W, Kang M, Wang J, Xu T, Xu M, Zhi L, Liu Q, Wang N, Zhou C. Efficacy and safety of KN046, a novel bispecific antibody against PD-L1 and CTLA-4, in patients with non-small cell lung cancer who failed platinum-based chemotherapy: a phase II study. Eur J Cancer. 2023 Sep;190:112936. doi: 10.1016/j.ejca.2023.05.024. Epub 2023 Jun 5. PMID 37393762
- [Derived] Song X, Xiong A, Wu F, Li X, Wang J, Jiang T, Chen P, Zhang X, Zhao Z, Liu H, Cheng L, Zhao C, Wang Z, Pan C, Cui X, Xu T, Luo H, Zhou C. Spatial multi-omics revealed the impact of tumor ecosystem heterogeneity on immunotherapy efficacy in patients with advanced non-small cell lung cancer treated with bispecific antibody. J Immunother Cancer. 2023 Feb;11(2):e006234. doi: 10.1136/jitc-2022-006234. PMID 36854570